CLINICAL TRIAL: NCT05972694
Title: The Effect of Grapes in Inflammatory Bowel Disease
Brief Title: Effect of Grapes in Inflammatory Bowel Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20230070
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: subjects will continue to consume their usual diet (excluding all grapes/berries) and consume 46g/d freeze-dried grape powder daily (consumed as 22.5g packets twice daily for 21 days. A stool and blood sample will be collected at the start and end of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Freeze-dried Grape powder intervention (Experimental): participants will be supplemented with 46g/d freeze-dried grape powder consumed as 22.5g packets twice daily for 21 days.
  Interventions: Dietary Supplement: Freeze dried grape powder

INTERVENTIONS:
Dietary Supplement: Freeze dried grape powder — 46g/d freeze-dried grape powder

SUMMARY:
The overall objective of this pilot intervention study is to determine the impact of grape powder (46g/day freeze dried whole grape powder provided by the California Table Grape Commission) on the gut microbiotacomposition in adult patients with the IBD subtype Crohn's disease (CD).

DETAILED DESCRIPTION:
This protocol is designed to investigate the effect of grape powder consumption in Inflammatory Bowel Disease (IBD), in particular how grape powder consumption (provided as 46g/day grape powder; equivalent to 1.5 cups fresh grapes) alters the gut microbiota (GM) composition in humans with IBD. The investigators will focus on studying IBD patients affected with CD as a proof of principle that could be tested later in other IBD subtype (ulcerative colitis or others specific surgical conditions).

The overall objective of this pilot intervention study is to determine the impact of grape powder (46g/day freeze dried whole grape powder provided by the California Table Grape Commission) on the GM composition in adult patients with the IBD subtype Crohn's disease (CD).

An 28 day pilot study in adult CD patients at the Digestive Health Institutes (DHI) of University Hospitals Cleveland Medical Center (UHCMC). table

Participation in this study will last for a maximum of 28 days and will consist of two phases. Phase I (baseline period - 7 days) where all grapes and berries will be removed from the diet, and Phase II (intervention period - 21 days) where participants will be supplemented with 46g/d freeze-dried grape powder consumed as 22.5g packets twice daily. The dose of 46g/day of grape powder is equivalent to 1.5 cups of grapes. Participants will be asked to avoid consumption of all other grapes/berries during phase II. The investigators will compare the before and after changes in gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Crohns disease. CD outpatients in remission
* Harvey Bradshaw-index in remission (<6 score)
* Capable of providing consent to participate.
* Able to complete daily surveys and take oral nutrition
* Able to record daily meal intake

Exclusion Criteria:

* Short bowel syndrome.
* Hospitalized patients.
* Individuals who lack consent capacity, including the mentally ill, prisoners, cognitively impaired participants, dementia patients.
* Known drug abuse.
* Known parasitic disease of the digestive system.
* Symptomatic intestinal stricture.
* Presence of an ostomy.
* Other conditions that would be a contraindication to consumption of the study diets or preclude the participant from completing the study.
* Well-founded doubt about the patients cooperation.
* Existing pregnancy or lactation.
* History of <1 natural bowel movements per day.
* Unable to access to technology that permits the daily completion of study related activities.
* Change in IBD medication within past 4 weeks.
* Body mass Index <16 kg/m or ≥35.
* Documented C.difficile colitis within four weeks of screening.
* Known berry or grape allergy
* No probiotic or antibiotic use for the previous 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
fecal microbiota composition | baseline (pre-intervention), immediately after the intervention
  16S microbiome

SECONDARY OUTCOMES:
fecal myleoperoxidase (MPO) | baseline (pre-intervention), immediately after the intervention
  fecal marker of inflammation
fecal calprotectin | baseline (pre-intervention), immediately after the intervention
  fecal marker of inflammation
C-reactive protein (CRP) | baseline (pre-intervention), immediately after the intervention
  blood marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Basson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: California Table Grape Commission — http://www.grapesfromcalifornia.com/